CLINICAL TRIAL: NCT01955928
Title: Internet-delivered CBT for Insomnia: Role of Sleep-related Cognitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Jaap Lancee, PhD, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UvA-2013-KP-3152
Record Dates: First submitted 2013-09-21; First posted 2013-10-08 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (2):
- Online Cognitive behavioral treatment for insomnia (Experimental): Online Cognitive behavioral treatment for insomnia
  Interventions: Behavioral: Online Cognitive behavioral treatment for insomnia
- Waiting-list (No Intervention): Waiting-list

INTERVENTIONS:
Behavioral: Online Cognitive behavioral treatment for insomnia
  Arms: Online Cognitive behavioral treatment for insomnia

SUMMARY:
The object of this study is to compare internet-delivered treatment for insomnia to a waiting-list. In this study participants are randomized to: 1) online cognitive-behavioral 2) waiting-list. Participants in the waiting-list condition receive treatment after the post-test. The interventions consist of: diary; psycho-education; relaxation exercises; stimulus control/sleep hygiene; sleep restriction; challenging the misconceptions about sleep; and paradoxical exercise. Adult persons with insomnia will be invited via a popular scientific website to fill out online questionnaires. Participants will fill out questionnaires and a dairy at baseline post-test, 3-month follow-up, and 6-month follow-up. In this study we are interested in sleep-related worry and daily complaints measured with a diary. We expect that the online intervention ameliorates both the sleep-related worry and the daily complaints. Furthermore, we expect that the sleep related worry mediates the effect of the intervention on sleep- and daily complaints.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia disorder according to DSM-5
* Sleep onset latency/wake after sleep onset > 30 minutes , three times or more a week
* Insomnia three months or longer
* Access to internet

Exclusion Criteria:

* Earlier cognitive behavioral treatment for insomnia
* Start other psychological treatment in the last 6 months
* Doing shift work
* Pregnancy or breast feeding
* Schizophrenia or psychosis
* Suicidal plans
* Sleep apnea
* drugs or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Daytime symptoms of sleep related worry measured with the APSQ | Change from baseline to post-test, 3-months, and 6-months follow-up
  Daytime symptoms of sleep related worry will be measured with a daily Anxiety and Pre-occupation about sleep questionnaire.
Daytime symptoms measured with diary consisting of the DASS-21 | Change from baseline to post-test, 3-months, and 6-months follow-up
  The daytime symptoms will be measured with the 7 items of the stress scale of the DASS-21

SECONDARY OUTCOMES:
Depression measured with the CES-D | Change from baseline to post-test, 3-months, and 6-months follow-up
Anxiety measured with the HADS-A | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related safety behaviors measured with the SRBQ | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related arousal measured with the Pre-arousal sleep scale | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related worry measured with the Anxiety and Pre-occupation about Sleep Scale | Change from baseline to post-test, 3-months, and 6-months follow-up
Repetitive thinking measured with the Dutch Perseverative Thinking Questionnaire | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related cognitions measured with the Dysfunctional Beliefs and Attitudes about sleep scale (DBAS) | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep medication usage per day measured with the sleep diary | Change from baseline to post-test, 3-months, and 6-months follow-up
sleep continuity (consisting of sleep latency, time awake after sleep onset, total sleep time) | Change from baseline to post-test, 3-months, and 6-months follow-up
  Sleep continuity is measured with a 7-day sleep diary based on the consensus sleep diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Psychology, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Result] Lancee J, Eisma MC, van Straten A, Kamphuis JH. Sleep-Related Safety Behaviors and Dysfunctional Beliefs Mediate the Efficacy of Online CBT for Insomnia: A Randomized Controlled Trial. Cogn Behav Ther. 2015;44(5):406-22. doi: 10.1080/16506073.2015.1026386. Epub 2015 May 27. PMID 26012890
- See also: General website about insomnia — http://www.insomnie.nl